CLINICAL TRIAL: NCT02375607
Title: Could Algometric Assessment be Effective to Adjust Postoperative Analgesic Requirement?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ziya Kaya, Associate Professor, MD, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 26/07/2011-195
Record Dates: First submitted 2015-02-10; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: Pain management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Algometer (Other): Algometer used patients
  Interventions: Device: Algometer

INTERVENTIONS:
Device: Algometer — Algometer performed patients
  Other Names: J-Tech Commander - Algometer

SUMMARY:
The purpose of this study is to determine the correlation between preoperative algometer score and the amount of postoperative analgesic consumption. The algometer score of the patients will be recorded in the preoperative period. In postoperative period, the analgesic consumption rate will record and compare with the algometer score.

DETAILED DESCRIPTION:
The aim of this study is to define the correlation between preoperative algometer score and the analgesic consumption rate. A total of 80 patients whose undergo septoplasty or septorhinoplasty will be included in this study. After preoperative examination, a positive pressure using algometer device will be performed until minimal pain is felt. In postoperative period, the amount of analgesic consumption of the patient will record and compare with the algometer score.

ELIGIBILITY:
Inclusion Criteria:

* Patients those undergo septoplasty or septorhinoplasty

Exclusion Criteria:

* Hypertension
* Diabetes mellitus type 1 or 2
* Continuous use of analgesics
* Patients whose do not accept to participate in the study
* Patients those reoperated for bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Algometer score | In one hour before the operation up to 3 years
  Score obtained from the Algometer device

SECONDARY OUTCOMES:
Analgesic consumption | In the first 24 hours after the operation up to 3 years
  The amount of analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: ZIYA KAYA, Assoc.Prof., Principal Investigator — Gaziosmanpasa University, Medical Faculty, Department of Anesthesiology and Reanimation
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Background] Hsu YW, Somma J, Hung YC, Tsai PS, Yang CH, Chen CC. Predicting postoperative pain by preoperative pressure pain assessment. Anesthesiology. 2005 Sep;103(3):613-8. doi: 10.1097/00000542-200509000-00026. PMID 16129988